CLINICAL TRIAL: NCT06147193
Title: Effects of Resistance Sprint Training With and Without Power Training on Sprint and Agility Performance in Football Players
Brief Title: Effects of Resistance Sprint Training With and Without Power Training on Sprint and Agility Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCRS/1021 Tehreem
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Resistance Sprint Training With and Without Power
Keywords: Agility Training; Football; Power Training; Resistance Sprint Training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power training Group (Active Comparator): with baseline intervention and power training interventions
  Interventions: Other: with baseline intervention and power training interventions
- Baseline Group (Other): baseline interventions and without power training interventions
  Interventions: Other: baseline interventions and without power training interventions

INTERVENTIONS:
Other: with baseline intervention and power training interventions — Group A (with power training ) was treated with
  * squats jump,
  * change of direction speed,
  * countermovement jump,
  * bench press,
  * Romanian deadlift
  * barbell squats,
  * resistance band sprints,
  * stair sprints
  * weighted sled pulls
  Arms: Power training Group
Other: baseline interventions and without power training interventions — Group B (without power training) was treated with
  * squats jump
  * change of direction speed
  * countermovement jump
  * barbell squats
  * resistance band sprints
  * stair sprints
  * Weighted sled pulls.
  Arms: Baseline Group

SUMMARY:
This study will be randomized clinical trial will be used to get expected outcomes. Hence under ethical consideration athletes of Pakistan football federation will go under the selection criteria and chosen voluntarily to participate in the study. Data will be collected with non-probability convenient sampling technique and 40 football players will be participated in this study. Participates will be divided into two groups with randomization process. 20 athletes will be in each group. Group A will be treated with squats jumps, change of direction speed, countermovement jump, bench press, Romanian deadlift and barbell squats, resistance band sprints, stair sprints and weighted sled pulls and Group B will be treated with squats jumps, change of direction speed, countermovement jump, resistance band sprints, stairs sprints and weighted sled pulls. These exercises will be given in 3 sets with 10 repetitions in each set. Pre and post interventions measures will be taken on 1st day and at 6th week there will be 3 sessions in a week. SPSS version 25 will be used to analyze the data.

DETAILED DESCRIPTION:
Football is a sport which is of high-intensity intermittent game that requires players to be physically capable of coping with high-intensity movements, having repeated changes of direction, sprints, and accelerations/decelerations, with complex and physically demanding technical different actions Developing and loading strength techniques in football come from knowledge of game performance and its specific components and limitation components. Most of the important factors in football are explosiveness activities such as changing direction, jumping, sprinting, and kicking. Working on these explosive performances have been found after strength training that improved the available force of muscular contraction in appropriate muscle groups. Vertical jump and sprint performances are interlinked with maximal muscular strength in football players and the heavy resistance training can also increase running economy and which ultimately increases the aerobic performance of the athlete

ELIGIBILITY:
Inclusion Criteria:

* Male football players
* Age 18- 40 years
* BMI 18.5-25
* Being volunteered to participate in study
* Being engaged in practice from past 6th month

Exclusion Criteria:

* Athlete with current substance abuse
* Individual diagnose with severe anxiety disorder and psychosis
* History of previous fracture from last 6 months
* Musculoskeletal disorders (sprains, strains, tendinopathies, stress fracture)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Resisted sprinting speeds at 10-30 m | Change from Baseline at 6 weeks
  The athlete sprints a distance of 10-30m while pushing or pulling against resistance. This resistance can be provided by various means, such as sled, resistance band, or a partner holding onto a harness worn by athlete. A study suggested that the magnitude of the correlation coefficient between speed-test results and match parameters was considered as small (0.1 ≤ r < 0.3), moderate (0.3 ≤ r < 0.5), large (0.5 ≤ r < 0.7), very large (0.7 ≤ r < 0.9), and nearly perfect (r ≥ 0.9)
Change of direction speed (COD) testing | Change from Baseline at 6 weeks
  This test consists of four 5-m sections marked with cones set at 100° angles. Three maximal attempts were performed with a 5-min rest interval between attempts. Starting from a standing position with the front foot placed 0.3 m behind the first pair of photocells i.e., starting line athletes ran and changed direction as quickly as possible until crossing the second pair of photocells placed 20 m from the starting line .A study suggests a near perfect correlation between the COD (r=0.92)
Squat jumps (SJ) | Change from Baseline at 6 weeks
  In the SJ, a static position with a 90° knee flexion angle was maintained for 2 seconds before every jump attempt. No preparatory movement was allowed and an experienced researcher visually inspected for proper technique. A study suggested that jumping tests had high correlation coefficients with the principal component (r = 0.76-0.87.
Countermovement Jump (CMJ) | Change from Baseline at 6 weeks
  In the CMJ, athletes were instructed to perform a downward movement followed by a complete extension of the lower limbs and were allowed to freely determine the amplitude of the countermovement to avoid changes in their jumping coordination pattern. Participants were instructed to assume the same body position at takeoff and landing on both squat and counter movement jumps) the CMJ tests had a high correlation coefficient with the principal component (r=0.76-0.87)
Horizontal Jump (HJ) | Change from Baseline at 6 weeks
  The athlete stands behind a line marked on the ground with feet slightly apart. A two-foot take-off and landing is used, with swinging of the arms and bending of the knees to provide forward drive. The subject attempts to jump as far as possible, landing on both feet without falling backwards. Three attempts are allowed a study suggested a Horizontal jump assessment(r=-0.7-0.86)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Ghafoor, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Combs B, Fazeli PL, Brown DA, Gallagher S, Jones A, Romeo B, Heaton K. Description of the Nature of Musculoskeletal Shoulder Injuries in a Cohort of Commercial Truck Drivers: A Retrospective Cross-Sectional Study. Workplace Health Saf. 2021 Aug;69(8):375-382. doi: 10.1177/2165079921990364. Epub 2021 Apr 13. PMID 33845688
- [Background] O'Brien L, Collins K, Amirabdollhian F. Exploring Sports Nutrition Knowledge in Elite Gaelic Footballers. Nutrients. 2021 Mar 26;13(4):1081. doi: 10.3390/nu13041081. PMID 33810237
- [Background] Hasan S, Kandasamy G, Alyahya D, Alonazi A, Jamal A, Unnikrishnan R, Muthusamy H, Iqbal A. Effect of Resisted Sprint and Plyometric Training on Lower Limb Functional Performance in Collegiate Male Football Players: A Randomised Control Trial. Int J Environ Res Public Health. 2021 Jun 22;18(13):6702. doi: 10.3390/ijerph18136702. PMID 34206346
- [Background] Gil S, Barroso R, Crivoi do Carmo E, Loturco I, Kobal R, Tricoli V, Ugrinowitsch C, Roschel H. Effects of resisted sprint training on sprinting ability and change of direction speed in professional soccer players. J Sports Sci. 2018 Sep;36(17):1923-1929. doi: 10.1080/02640414.2018.1426346. Epub 2018 Jan 15. PMID 29334309
- [Background] Pacholek M, Zemkova E. Effect of Two Strength Training Models on Muscle Power and Strength in Elite Women's Football Players. Sports (Basel). 2020 Mar 30;8(4):42. doi: 10.3390/sports8040042. PMID 32235425
- [Background] Altmann S, Ringhof S, Neumann R, Woll A, Rumpf MC. Validity and reliability of speed tests used in soccer: A systematic review. PLoS One. 2019 Aug 14;14(8):e0220982. doi: 10.1371/journal.pone.0220982. eCollection 2019. PMID 31412057
- [Background] Beato M, Bianchi M, Coratella G, Merlini M, Drust B. Effects of Plyometric and Directional Training on Speed and Jump Performance in Elite Youth Soccer Players. J Strength Cond Res. 2018 Feb;32(2):289-296. doi: 10.1519/JSC.0000000000002371. PMID 29176387
- [Background] Van Hooren B, Zolotarjova J. The Difference Between Countermovement and Squat Jump Performances: A Review of Underlying Mechanisms With Practical Applications. J Strength Cond Res. 2017 Jul;31(7):2011-2020. doi: 10.1519/JSC.0000000000001913. PMID 28640774
- [Background] Markovic G, Dizdar D, Jukic I, Cardinale M. Reliability and factorial validity of squat and countermovement jump tests. J Strength Cond Res. 2004 Aug;18(3):551-5. doi: 10.1519/1533-4287(2004)182.0.CO;2. PMID 15320660